CLINICAL TRIAL: NCT06923891
Title: An Open-Label Study to Evaluate the Efficacy and Tolerability of Xanomeline/Trospium In First Episode/Early Phase Schizophrenia Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Vanguard Research Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEP Cobenfy
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Xanomeline/Trospium (Active Comparator): Cobenfy
  Interventions: Drug: Xanomeline/Trospium

INTERVENTIONS:
Drug: Xanomeline/Trospium — Xanomeline/Trospium (titrated dose)
  Other Names: Cobenfy

SUMMARY:
This is an open label study of the treatment satisfaction, efficacy and tolerability of xanomeline/ trospium in a population of 172 participants diagnosed with schizophrenia in the early phase of illness. Participants will be followed for 24 weeks with scheduled assessments conducted by centralized raters, local mental health professionals and self-assessments completed by patients. Recruitment will be based on insufficient efficacy of previous antipsychotic or due to dissatisfaction with treatment as a result of unacceptable side effects on previous antipsychotic/patient choice, with approximately 50% for each enrollment criteria. Participants who present with both insufficient efficacy and unacceptable side effects will be considered as belonging to the insufficient efficacy subgroup. Treatment and assessments will be identical for the 2 groups. Primary outcome for participants enrolled will be improvement in overall treatment satisfaction as measured by the MSQ.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is aged 18-40 years, inclusive, at time of signing the ICF
2. Participant has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 (American Psychiatric Association 2013) criteria and confirmed by Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorder Studies (MINI) version 7.0.2.
3. Participant Scores MSQ ≤3 for the Medication Satisfaction Questionnaire (MSQ)
4. Within 5 years of first antipsychotic treatment for psychosis at time of signing ICF
5. Clinical reason to seek a change in antipsychotic treatment due to psychosis symptom severity, it is clinically appropriate for the participant to seek a change in antipsychotic treatment due to psychosis symptom severity, adverse effects, both, or overall patient judgement/choice.
6. Symptom Severity Criteria:

   1. Clinical reasons include Positive and Negative Syndrome Scale (PANSS) total score of ≤ 120 at screening if participant is experiencing inefficacy from current antipsychotic treatment and
   2. A score of ≥ 4 (moderate or greater) for ≥ 1 of the following PANSS Positive Subscale (P) items: i. Item 1 (P1; delusions), ii. Item 2 (P2; conceptual disorganization), iii. Item 3 (P3; hallucinatory behavior), iv. Item 6 (P6; suspiciousness/persecution) and
   3. A Clinical Global Impressions-Severity scale (CGI-S) score of ≥ 4 at screening and baseline visits.

   OR
7. Adverse Event or Overall Patient Choice Criteria:

   1. A score of <4 for all the following PANSS Positive Subscale (P) items: i. Item 1 (P1; delusions), ii. Item 2 (P2; conceptual disorganization), iii. Item 3 (P3; hallucinatory behavior), iv. Item 6 (P6; suspiciousness/persecution)
   2. Participant Scores MSQ ≤3 for the Medication Satisfaction Questionnaire (MSQ)Clinical reason to seek a change in antipsychotic treatment due to adverse effects or overall patient judgement/choice.
8. Upon screening, the treatment plan is for outpatient level of care. Transition to inpatient level of care after enrollment does not exclude the patient from participating in the study
9. Participant is taking an antipsychotic (AP) and the AP regimen has been stable for at least 8 weeks with at least the last 4 weeks on the same dose (i.e., untreated patients or patients receiving antipsychotic polypharmacy are excluded) prior to Screening. Participants are permitted to remain on non-prohibited (see, Exclusion Criterion, and Section 9) psychotropic medications (that are not secondary AP treatments) other than the primary pre-switch AP that have been part of their ongoing treatment regimen.

   a. Anticholinergic drugs (e.g., benztropine) are allowed at baseline but need to be washed out during cross titration within 1 week after initiating xanomeline/trospium.
10. Subject can provide informed consent. A signed informed consent form must be provided before any study assessments are performed. Subject must be fluent (oral and written) in English to consent. Female participants must be willing and capable to use birth control throughout the time of the trial as defined in Section 3.1.3

Exclusion Criteria:

1. Any DSM-5 disorder other than schizophrenia within 6 months before screening (confirmed using MINI version 7.0.2 at screening) requiring clinical attention.
2. Active substance or alcohol abuse or dependence in the past 6 months (cannabis use is allowed if not fulfilling abuse criteria)
3. Urine toxicology screen is positive for phencyclidine, amphetamines, opiates, cocaine, or alcohol (clinically significant alcohol use in the opinion of the Investigator)
4. Developmental disorder or intellectual disability
5. History of serious suicide attempt within the past 6 months
6. Risk of suicidal behavior as determined by the Investigator's clinical assessment. Lifetime history of clinically significant head trauma, or current history of other acute or serious medical condition or
7. History or presence of clinically significant cardiovascular (eg, untreated or unstable hypertension, clinically significant tachycardia), pulmonary, renal, hematologic, gastrointestinal ([GI] e.g., obstructive disorders [including conditions that may decrease GI motility, such as ulcerative colitis, intestinal atony, and myasthenia gravis], endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results.
8. Active biliary disease (eg, symptomatic gallstones). Participants with other biliary histories are eligible and should be discussed with the medical monitor
9. History or high risk of urinary retention, gastric retention,
10. Untreated narrow-angle glaucoma
11. An estimated glomerular filtration rate (eGFR) of < 60 mL/min at the screening visit.
12. Elevations in hepatic transaminases at screening ≥ 3× ULN for ALT and AST and/or ≥ 2× ULN for total bilirubin
13. History of hypersensitivity or prior exposure to xanomeline/trospium or trospium chloride
14. History of any significant drug allergy (such as anaphylaxis or hepatotoxicity).
15. Intellectual disability or autism spectrum disorder (by history)
16. Active substance dependence within the past 3 months (except for tobacco and cannabis)
17. Participant has a history of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 6 weeks at an adequate dose per the label), based on TRIPP guidelines (Howes, et al 2017).
18. Participant is on or has history of clozapine treatment
19. Participant is on≥ 2 antipsychotics at baseline
20. Participant has received a long-acting injectable antipsychotic within one injection cycle for that formulation at the time of baseline (i.e., cycles are defined by the interval in which the LAI is administered. If it is a monthly administration, then the exclusion is for one month since the last LAI administration).
21. Participant is receiving other psychotropic medications other than the antipsychotic to be switched, for psychiatric and neurological drugs with Anticholinergic Risk Scale (ARS) scores >1 (tricyclic antidepressants, paroxetine, antispasmodics, antihistamines with anticholinergic properties).
22. Active biliary disease (eg, symptomatic gallstones). Participants with other biliary histories are eligible and should be discussed with the medical monitor
23. Pregnancy, breastfeeding or less than 3 months postpartum or intent to get pregnant within the next 6 months
24. Participants with any of the following:

    1. history of bladder stones
    2. history of recurrent urinary tract infections
25. History of unstable hypertension or tachycardia as evidenced by:

    1. Blood pressure of ≥ 160/100 mmHg (seated measures) at screening
    2. Heart rate of ≥ 110 bpm (seated measures) at screening
26. Clinically significant abnormal finding on the physical examination, medical history, or clinical laboratory results at Screening
27. Current participation in another clinical trial, or participation in another clinical study in which the participant received an experimental or investigational drug agent within 3 months prior to screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-04-16 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Medication Satisfaction Questionnaire (MSQ) | 12 weeks
  Change in total MSQ from baseline to week 12

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 12 weeks
  PANSS total score from baseline to week 12
Clinical Global Impression - Severity Scale (CGI-S) | 12 weeks
  CGI-S score from baseline to week 12
Treatment Satisfaction Questionnaire for Medication (TSQM) | 12 weeks
  Change in TSMQ global satisfaction from baseline to week 12
Personal and social performance scale (PSP) | 12 weeks
  Personal and social performance scale (PSP) scores from baseline to week 12
All cause discontinuation | 12 weeks
  All-cause and specific-cause discontinuation by week 12
Merck Adherence Estimator | 12 weeks
  Adherence (Merck Adherence Estimator), from baseline to week 12
Adverse Effects | 12 weeks
  Incidence of adverse effects for overall study period to and of safety follow up by week 12
Columbia Suicidal Severity Rating Scale (C-SSRS) | 12 weeks
  Columbia Suicidal Severity Rating Scale (C-SSRS) by week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Richmond, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Howes OD, McCutcheon R, Agid O, de Bartolomeis A, van Beveren NJ, Birnbaum ML, Bloomfield MA, Bressan RA, Buchanan RW, Carpenter WT, Castle DJ, Citrome L, Daskalakis ZJ, Davidson M, Drake RJ, Dursun S, Ebdrup BH, Elkis H, Falkai P, Fleischacker WW, Gadelha A, Gaughran F, Glenthoj BY, Graff-Guerrero A, Hallak JE, Honer WG, Kennedy J, Kinon BJ, Lawrie SM, Lee J, Leweke FM, MacCabe JH, McNabb CB, Meltzer H, Moller HJ, Nakajima S, Pantelis C, Reis Marques T, Remington G, Rossell SL, Russell BR, Siu CO, Suzuki T, Sommer IE, Taylor D, Thomas N, Ucok A, Umbricht D, Walters JT, Kane J, Correll CU. Treatment-Resistant Schizophrenia: Treatment Response and Resistance in Psychosis (TRRIP) Working Group Consensus Guidelines on Diagnosis and Terminology. Am J Psychiatry. 2017 Mar 1;174(3):216-229. doi: 10.1176/appi.ajp.2016.16050503. Epub 2016 Dec 6. PMID 27919182
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27919182/